CLINICAL TRIAL: NCT00807612
Title: A Phase 1b/2 Study of AMG 479 in Combination With Paclitaxel and Carboplatin for the First-Line Treatment of Advanced Squamous Non-Small Cell Lung Cancer
Brief Title: QUILT-2.017: Phase 1b/2 Study of AMG 479 in Combination With Paclitaxel and Carboplatin for 1st Line Treatment of Advanced Squamous Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was closed due to administrative decision
Sponsor: NantCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20080257; QUILT-2.017 (Other: NantCell, Inc.)
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Advanced Squamous Non-Small Cell Lung Cancer
Keywords: AMG 479; IGF-1R; Apoptosis; Monoclonal Antibody; Advanced Squamous Non-Small Cell Lung Cancer; antibody 1st-line
MeSH Terms: conditions — Insulin-Like Growth Factor I, Resistance To | interventions — ganitumab; Carboplatin; Paclitaxel

ARMS (3):
- Part 1 Cohort 1 (Experimental): AMG 479 at 18 mg/kg in combination with paclitaxel/carboplatin for 4 to 6 cycles followed by AMG 479 at 18 mg/kg monotherapy for 24 months from study day 1
  Interventions: Biological: AMG 479; Drug: Carboplatin; Drug: Paclitaxel
- Part 1 Cohort 2 (Experimental): AMG 479 at 12 mg/kg in combination with paclitaxel/carboplatin for 4 to 6 cycles followed by AMG 479 at 12 mg/kg monotherapy for 24 months from study day 1
  Interventions: Biological: AMG 479; Drug: Carboplatin; Drug: Paclitaxel
- Part 2 (Experimental): AMG 479 in combination with paclitaxel/carboplatin for 4 to 6 cycles followed by AMG 479 monotherapy for 24 months from study day 1
  (AMG 479 dose in Part 2 will be the final AMG 479 dose from Part 1)
  Interventions: Drug: Carboplatin; Biological: AMG 479; Drug: Paclitaxel

INTERVENTIONS:
Biological: AMG 479 — AMG 479 at 12 mg/kg IV in combination with chemotherapy Day 1 of cycle 1 to 6 (except for subjects being evaluated by intensive PK who will be administered AMG 479 on day 2 of cycle 1 and then day 1 of every cycle thereafter) followed by AMG 479 at 12 mg/kg IV monotherapy for up to 24 months from study day 1
  Arms: Part 1 Cohort 2
Biological: AMG 479 — AMG 479 at 18mg/kg IV in combination with chemotherapy Day 1 of cycle 1 to 6 (except for subjects being evaluated by intensive PK who will be administered AMG 479 on Day 2 of cycle 1 and then day 1 of every cycle thereafter) followed by AMG 479 at 18 mg/kg IV monotherapy for up to 24 months from day 1
  Arms: Part 1 Cohort 1
Drug: Carboplatin — Carboplatin (AUC 6) IV infusion over 30 (± 10) minutes according to institutional guidelines Day 1 of Cycle 1 to 6
Biological: AMG 479 — AMG 479 IV in combination with chemotherapy on day 1 of every 3 week cycle for 4 to 6 cycles, followed by AMG 479 IV monotherapy for up to 24 months from study day 1. The AMG 479 dose to be used will be the final AMG 479 dose explored from Part 1
  Arms: Part 2
Drug: Paclitaxel — Paclitaxel at 200 mg/m2 IV infusion over 3 hours (± 30 minutes) according to institutional guidelines Day 1 of Cycle 1 to 6

SUMMARY:
This is a global, multicenter, 2-part, open-label phase 1b and single-arm phase 2 study designed to evaluate the safety and efficacy of AMG 479 in combination with paclitaxel and carboplatin for the first-line treatment of advanced squamous non-small cell lung carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced squamous NSCLC
* Measurable disease as defined per modified RECIST criteria
* ECOG performance status of 0 or 1
* ≥18 years old
* Adequate glycemic function, for subjects with known diabetes

Exclusion Criteria:

* Untreated or symptomatic central nervous system (CNS) metastases
* Prior anti-cancer therapy as follows: Any prior chemotherapy for squamous NSCLC; Any prior adjuvant or neoadjuvant chemotherapy for squamous NSCLC; Any prior chemoradiation for squamous NSCLC; Central (chest) radiation therapy ≤ 28 days prior to enrollment, radiation therapy for peripheral lesions≤14 days prior to enrollment for squamous NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (12):
- United States (12):
  - Research Site, Fayetteville, Arkansas
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Lafayette, Indiana
  - Research Site, New Albany, Indiana
  - Research Site, Paducah, Kentucky
  - Research Site, St Louis, Missouri
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Madison, Wisconsin

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Primary for discontinuing study 1 subject documented "completed" taken from "end-of-study" page of the CRF site entered ("end of study" defined all subjects that completed 60-day follow-up visit, death, 26 months post final subject randomization, whichever earlier). Based on the date of subject's end-of-study visit, primary reason likely the subject discontinued study to sponsor's early closing of the study. Part 1 and 2 were analyzed together because the same dose was given in both parts.
Groups:
- Ganitumab 18 mg/kg + Paclitaxel/Carboplatin: AMG 479 at 18 mg/kg in combination with paclitaxel/carboplatin for 4 to 6 cycles followed by AMG 479 at 18 mg/kg monotherapy for 24 months from study day 1
  AMG 479: AMG 479 at 18mg/kg IV in combination with chemotherapy Day 1 of cycle 1 to 6 (except for subjects being evaluated by intensive PK who will be administered AMG 479 on Day 2 of cycle 1 and then day 1 of every cycle thereafter) followed by AMG 479 at 18 mg/kg IV monotherapy for up to 24 months from day 1
  Carboplatin: Carboplatin (AUC 6) IV infusion over 30 (± 10) minutes according to institutional guidelines Day 1 of Cycle 1 to 6
  Paclitaxel: Paclitaxel at 200 mg/m2 IV infusion over 3 hours (± 30 minutes) according to institutional guidelines Day 1 of Cycle 1 to 6
Period: Overall Study
Arm/Group | Ganitumab 18 mg/kg + Paclitaxel/Carboplatin
Started | 15
Completed | 1
Not Completed | 14
Not completed — Death | 8
Not completed — Study early termination | 5
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 1 Subject completed the study and 14 subjects discontinued the study
Arm/Group | Ganitumab 18 mg/kg + Paclitaxel/Carboplatin
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Dose Limiting Toxicities
Description: DLTs were defined as grade 3 or higher hematological or nonhematological toxicities that, in the opinion of the investigator, were related to ganitumab or the combination of ganitumab and paclitaxel or carboplatin during this period. These did not include fatigue, nausea, diarrhea, vomiting, hyperglycemia, neutropenia, thrombocytopenia, anemia, lymphopenia, alopecia, increased ALT or AST, or pulmonary embolism unless they met certain criteria.
Time Frame: Part 1 only up to 21 days
Population: Dose-limiting-toxicity-evaluable subjects were defined as those who had received 1 dose of ganitumab in combination with paclitaxel and carboplatin and had completed 1 cycle (21 days) of study treatment or experienced a DLT related to ganitumab or the combination of ganitumab and paclitaxel/carboplatin during the first cycle (21 days) of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 479 18 mg/kg + Paclitaxel/Carboplatin
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Part 2: Objective Response Rate
Description: Part 2: Objective Response Rate as per modified RECIST criteria by investigator review Objective response was defined as a tumor response assessment of either complete response or partial response per modified Response Evaluation Criteria in Solid Tumors [RECIST] and was determined only for subjects with measurable disease at baseline. Per RECIST: a complete response is the disappearance of all target lesions; a partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From start of treatment up to approximately 16 months
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | AMG 479 18 mg/kg + Paclitaxel/Carboplatin
Number analyzed (Participants) | 15
percentage of participants | 27 [12 to 46]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events were assessed using CTCAE v 3.0
Time Frame: 30 days after last dose, up to 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 479 18 mg/kg + Paclitaxel/Carboplatin
Number analyzed (Participants) | 14
Participants | 14

4. Secondary Outcome: Number of Participants With Anti-AMG 479 Antibody Formation
Time Frame: From start of treatment up to approximately 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | AMG 479 18 mg/kg + Paclitaxel/Carboplatin
Number analyzed (Participants) | 15
Participants
  Total binding antibody incidence | 3
  neutralizing antibody incidence | 0

5. Secondary Outcome: Progression Free Survival
Description: PFS was defined as the time from study day 1 to the first observation of disease progression per investigator review (as classified by modified RECIST or death due to any cause, or censoring. Disease progression per RECIST is defined as at least a 20% increase in the sum of diameters of target lesions in reference to the smallest sum on study and an absolute increase of at least 5 mm; the appearance of any new lesions is also considered progression.
Time Frame: From start of treatment up to approximately 16 months
Measure: Median (80% Confidence Interval); unit: weeks
Arm/Group | AMG 479 18 mg/kg + Paclitaxel/Carboplatin
Number analyzed (Participants) | 15
weeks | 20.0 [14.1 to 23.7]

6. Secondary Outcome: Time to Progression and Duration of Response
Description: Time to Progression (TTP) is defined as the time from Day 1 to the first observation of disease progression (per modified RECIST). Disease progression per RECIST is defined as at least a 20% increase in the sum of diameters of target lesions in reference to the smallest sum on study and an absolute increase of at least 5 mm; the appearance of any new lesions is also considered progression. DOR was the time from the first observation of an objective response to the subsequent time of disease progression (per modified RECIST or clinical progression, whichever came first) or death due to any cause. Objective response = a tumor response assessment of either complete response or partial response per modified Response Evaluation Criteria in Solid Tumors [RECIST]. Per RECIST: a complete response is the disappearance of all target lesions; a partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From start of treatment up to approximately 16 months
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | AMG 479 18 mg/kg + Paclitaxel/Carboplatin
Number analyzed (Participants) | 15
Weeks
  Time to Progression | NA [NA to NA] — Median and confidence intervals are not available due to insufficient number of subjects with events.
  Duration of Response | NA [NA to NA] — Median and confidence intervals are not available due to insufficient number of subjects with events.

ADVERSE EVENTS:
Time Frame: 30 days after last dose, up to 5 months
Description: Safety analysis population was used for adverse events (only subjects with at least one dose of study drug). Mortality was calculated on all enrolled subjects.
Arm/Group | Ganitumab 18 mg/kg + Paclitaxel/Carboplatin
All-Cause Mortality (participants affected / at risk) | 8/15
Serious Adverse Events (participants affected / at risk) | 7/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganitumab 18 mg/kg + Paclitaxel/Carboplatin (N=14)
Pneumonia (Infections and infestations) | 3
Clostridial Infection (Infections and infestations) | 1
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tachycardia (Cardiac disorders) | 1
Asthenia (General disorders) | 1
Blood Amylase Increased (Investigations) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ganitumab 18 mg/kg + Paclitaxel/Carboplatin (N=14)
Nausea (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 12
Asthenia (General disorders) | 3
Oedema Peripheral (General disorders) | 3
Chills (General disorders) | 2
Pyrexia (General disorders) | 2
Adverse Drug Reaction (General disorders) | 1
Chest Pain (General disorders) | 1
Infusion Related Reaction (General disorders) | 1
Oedema (General disorders) | 1
Pain (General disorders) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Dysgeusia (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 5
Peripheral Sensory Neuropathy (Nervous system disorders) | 5
Headache (Nervous system disorders) | 3
Peripheral Motor Neuropathy (Nervous system disorders) | 3
Aphasia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Neuropathy Peripheral (Nervous system disorders) | 1
Restless Legs Syndrome (Nervous system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash Follicular (Skin and subcutaneous tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Pneumonia (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Lung Infection (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2
Bacteraemia (Infections and infestations) | 1
Clostridial Infection (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Confusional State (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Alanine Aminotransferase Increased (Investigations) | 2
Aspartate Aminotransferase Increased (Investigations) | 1
Blood Amylase Increased (Investigations) | 1
Blood Creatinine Increased (Investigations) | 1
International Normalised Ratio Increased (Investigations) | 1
Weight Decreased (Investigations) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Deep Vein Thrombosis (Vascular disorders) | 1
Orthostatic Hypotension (Vascular disorders) | 1
Superior Vena Caval Occlusion (Vascular disorders) | 1
Supraventricular Tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Eye Swelling (Eye disorders) | 1
Photopsia (Eye disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Ankle Fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pollakiuria (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Galactorrhoea (Reproductive system and breast disorders) | 1

LIMITATIONS AND CAVEATS:
There was a small number of subjects enrolled (15, only 14 treated) compared to the planned sample size (up to 52) and small number of responses/events occurring which could introduce bias in interpretation of the results and potentially misleading conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-08-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT00807612/Prot_SAP_000.pdf